CLINICAL TRIAL: NCT00163787
Title: Clinical Identification of Increased Fall Risk Early After Unilateral Transtibial Amputation
Brief Title: Clinical Identification of Fall Risk Early After Unilateral Transtibial Amputation
Status: Completed | Type: Observational
Sponsor: Bayside Health (Other Government)
Collaborators: Austin Health (Other Government)
Other Study IDs: 79/03
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-09

CONDITIONS: Amputation
Keywords: mobility; falls; activity level
MeSH Terms: interventions — Outcome Assessment, Health Care; Self Report

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

INTERVENTIONS:
Behavioral: outcome measures and self report

SUMMARY:
All participants attend for two testing sessions at either Royal Talbot Rehabilitation Centre or the centre where they received inpatient physiotherapy services.

All participants will be tested at discharge and at six months post discharge. Personnel used to score and administer the balance tests at six months will be blinded to pre-test scores, subject background, as well as, mobility and fall history in the six months post discharge.

At discharge participants will perform two successful Four Square Step Tests (FSST, and will be videotaped performing the Timed Up and Go Test (TUGT. The turn measure will be scored from this TUGT. Participants will also complete the Locomotor Capabilities index (LCI).

At the six-month test participants repeat balance and mobility tests and LCI, as well as being interviewed to ascertain fall history since discharge.

DETAILED DESCRIPTION:
Subjects:

All unilateral trans-tibial amputees with prosthesis at discharge, who are over 18 years of age, willing to participate and give informed consent. Subjects will be excluded if visually unable to perform tests, cognitively unable to follow testing procedures or being discharged into supported accommodation.

Identify scores for unilateral trans-tibial amputees for; FSST, TUGT and turn measure items: (1) steps, (2) time and (3) steadiness & fluency of movement.

Evaluate the validity, predictive value, sensitivity & specificity of the balance and mobility measures for falls and community ambulation with trans-tibial amputees.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years unilateral transtibial amputee

Exclusion Criteria:

* visually unable to perform tests cognitively unable to perform tests unable to provide informed consent not being discharged into supported accommodation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-06; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Mr Dite, MAppSci, Principal Investigator — Austin Health Royal Talbot Rehabilitation Centre
Locations (1):
- Austin Health Royal Talbot Rehabilitation Centre, Melbourne, Victoria, Australia